CLINICAL TRIAL: NCT00894946
Title: The in Vitro Fertilisation - Lipiodol Uterine Bathing Effect Study
Brief Title: The In Vitro Fertilization - Lipiodol Uterine Bathing Effect Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Associate Professor Neil Johnson, University of Auckland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVF-LUBE
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Endometriosis; In Vitro Fertilization Implantation Failure
Keywords: recurrent IVF implantation failure
MeSH Terms: conditions — Endometriosis | interventions — Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recurrent IVF implantation failure (Experimental)
  Interventions: Procedure: Lipiodol + IVF; Procedure: IVF
- Endometriosis (Experimental)
  Interventions: Procedure: Lipiodol + IVF; Procedure: IVF

INTERVENTIONS:
Procedure: Lipiodol + IVF — IVF preceded by lipiodol
Procedure: IVF — IVF alone

SUMMARY:
The hypothesis of this study is that Lipiodol uterine bathing improves the success rate of in vitro fertilization (IVF) for women with endometriosis or recurrent IVF implantation failure.

ELIGIBILITY:
Inclusion Criteria:

* 12 or more months infertility
* Age 18 to 39
* Endometriosis or recurrent IVF implantation failure
* Patent fallopian tubes

Exclusion Criteria:

* Iodine allergy
* Blocked fallopian tube or tubes

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2009-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Live birth | 12 months post-randomization

SECONDARY OUTCOMES:
Clinical pregnancy | 3 months post-randomization
Adverse events | 3 & 12 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Neil Johnson, MD, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- University of Auckland, Auckland, New Zealand